CLINICAL TRIAL: NCT02790541
Title: Changes in Blood Flow and Angiogenesis Induced in the Elderly by Hyperbaric Oxygen Therapy
Brief Title: Angiogenesis Induced in the Elderly by Hyperbaric Oxygen Therapy
Acronym: ANGIOHBOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, MD, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0172-15-ASF
Record Dates: First submitted 2016-05-03; First posted 2016-06-06 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Aging
Keywords: aging; HBOT; reverse; angiogenesis; elderly; mitochohndria
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Hyperbaric Oxygen Therapy: 3 months of treatment consisting of 60 daily sessions, 90 minutes of 100% oxygen at pressure of 2 ATA each, five days a week
  Interventions: Device: Hyperbaric Oxygen Therapy
- Control/Crossover (Other): Hyperbaric Oxygen Therapy: 3 months control period (no treatment) followed by 3 months of treatment consisting of 60 daily sessions, 90 minutes of 100% oxygen at pressure of 2 ATA each, five days a week
  Interventions: Device: Hyperbaric Oxygen Therapy

INTERVENTIONS:
Device: Hyperbaric Oxygen Therapy — 60 daily sessions, 90 minutes of 100% oxygen at pressure of 2 ATA each, five days a week for 3 months.
  Other Names: HBOT

SUMMARY:
Recent studies show preliminary evidence of HBOT therapeutic effects on angiogenesis, increased tissue blood flow and oxygenation correlated with tissue function.

Our primary hypothesis is that HBOT will have beneficial effects on the above mentioned organs associated with aging-related malfunctions due to restored mitochondrial function, mobilization of stem cells and induction of angiogenesis.

DETAILED DESCRIPTION:
The paradigm The accumulation of damage to molecules, cells and tissues over a lifetime that contributes to aging eventually leads to frailty and malfunction. The past decade has seen fundamental advances in our understanding of the aging process and raised optimism that interventions to slow ageing may be on the horizon. The aging process is linked to energy deficit due to tissue hypoxia and mitochondria dysfunction.

* Mitochondria dysfunction- Mitochondria are the primary generator of energy by means of ATP synthesis and their dysfunction leads to cellular function decline and degenerative changes. In addition, mitochondria dysfunction in stem cells decreases the capabilities for tissue regeneration.
* Tissue hypoxia- Atherosclerosis is a chronic inflammatory response that damages arterial blood vessels. It begins in childhood and progresses throughout life. A vicious cycle occurs as mitochondrial dysfunction accelerates atherosclerosis and the waning of microvasculature, resulting in decrease blood supply and ensuing relative tissue hypoxia. The decrease oxygen supply to the mitochondria further exacerbates mitochondrial dysfunction.

Hyperbaric oxygen can increase the partial pressure of dissolved (non-hemoglobin-bound) oxygen 20-30 fold and produce two main effects. First, it can eliminate the relative tissue hypoxia induced by atherosclerosis. Second, because mitochondria function is directly influenced by the partial pressure of dissolved oxygen, hyperbaric oxygen can amend mitochondrial dysfunction. Thus, the investigators suggest hyperbaric oxygen as a novel method for breaking the vicious cycle of degeneration and perhaps even for reversing the aging process.

The study is designed as a prospective crossover study aiming to evaluate the therapeutic effects of HBOT on the Brain, Cardiovascular and Immune system, Skin, Erectile (sexual functions), liver and Kidneys, of aging population.

After signing an informed consent form, patients will be invited for baseline evaluations. All patients would be evaluated 3 times - at baseline, after 3 months of follow up, and after additional 3 months of HBOT protocol. The evaluation will include cognitive assessment, questionnaires, MRI scans, blood tests and skin photograph and biopsy. In addition, blood tests will be drawn before and after the 20th, 40th and the 60th sessions for stem cells and mitochondria tests.

Patients will receive 60 daily sessions, 5 days/week, 90 minutes each with 5 minutes air break every 30 minutes, 100% oxygen at 2 ATA.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 65 years
* Capability to sign informed consent.
* No cardiac or cerebrovascular ischemia previous events one year prior to inclusion.

Exclusion Criteria:

* Previous treatment with HBOT for any other reason during the last 3 months prior to inclusion.
* Any history of malignancy during the last year prior to inclusion.
* Severe cognitive decline (MMSA<17)
* Severe chronic renal failure (GFR <30)
* Uncontrolled diabetes mellitus (HbA1C>8, fasting glucose>200)
* Immunosuppressant from any reason
* Contraindications to perform MRI: claustrophobia, allergy to gadolinium, foreign bodies, pacemaker, etc.
* Active Smoking.
* Pulmonary diseases such as severe emphysema, moderate-severe obstructive disease.
* Medical conditions deemed by the investigator to make the patient ineligible for protocol investigations.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-12; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Angiogenesis in brain MRI at 3 and 6 months | at baseline, 3 and 6 months
  imaging will be performed for evaluation of brain changes and angiogenesis processs using MRI perfusion (DSC)
Change from baseline of general cognitive functions index at 3 and 6 months | at baseline, 3 and 6 months
  Patients' cognitive functions will be assessed by Neurotrax computerized cognitive tests to generate the general cognitive index
Change from baseline of exercise VO2 MAX at 3 and 6 months | at baseline, 3 and 6 months
  Using a standard exercise test which includes gas analysis, the change in VO2 maxs will be assessed 3 and 6 months compared to baseline

SECONDARY OUTCOMES:
Change in number of circulating stem cells (CD34) at 3 and 6 months | at baseline, 3 and 6 months
  Blood samples will be drawn for measurements of CD34 stem cells number analyzed by FACS.
Change from baseline of proteinuria at 3 and 6 months | at baseline, 3 and 6 months
  24-hours urine will be collected from all patients for evaluation of proteinuria
Change from baseline of Methacetin breath test at 3 and 6 months | at baseline, 3 and 6 months
  All patients will undergo Methacetin breath test. Voltile CO2 levels will be compared to evaluate changes in liver function.
Change from baseline in bone density at 3 and 6 months | at baseline, 3 and 6 months
  All patients will undergo Dual-energy X-ray absorptiometry to evaluate the change bone density changes
Change from baseline in quality of life measured by SF-36 form at 3 and 6 months | at baseline, 3 and 6 months
  All patients will fill SF-36 questionnaire to evaluate the change in quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Asaf Harofeh Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hadanny A, Sasson E, Copel L, Daniel-Kotovsky M, Yaakobi E, Lang E, Fishlev G, Polak N, Friedman M, Doenyas K, Finci S, Zemel Y, Bechor Y, Efrati S. Physical enhancement of older adults using hyperbaric oxygen: a randomized controlled trial. BMC Geriatr. 2024 Jul 3;24(1):572. doi: 10.1186/s12877-024-05146-3. PMID 38961397